CLINICAL TRIAL: NCT00622193
Title: A Randomized, Double-Blind, Placebo-Controlled, Multicenter Phase II Anamorelin HCl Dose Range Study to Evaluate the Safety and Efficacy of Anamorelin HCl in Patients With NSCLC
Brief Title: Dose Range Study of Anamorelin in Patients With Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Helsinn Therapeutics (U.S.), Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ST-ANAM-207
Record Dates: First submitted 2008-02-12; First posted 2008-02-22 (Estimated); Last update posted 2017-04-14 (Actual); Status verified 2017-04

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 Active 50 mg (Experimental)
  Interventions: Drug: anamorelin HCl
- 2 Active 100 mg (Experimental)
  Interventions: Drug: anamorelin HCl
- 3 Placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: anamorelin HCl — 50 mg tablet
  Other Names: ST-1291
  Arms: 1 Active 50 mg
Drug: anamorelin HCl — 100 mg tablet
  Other Names: ST-1291
  Arms: 2 Active 100 mg
Drug: placebo — placebo tablet
  Arms: 3 Placebo

SUMMARY:
The purpose of this study is to evaluate doses of anamorelin for safety and efficacy in patients with non-small cell lung cancer.

DETAILED DESCRIPTION:
Cancer cachexia is a devastating, often late-stage complication of an underlying malignancy. Despite the significant importance of cancer-related cachexia, treatments are lacking and there are no products approved for this indication. Anamorelin HCl, by virtue of its ghrelin agonist activity, may serve a role in the treatment of cancer cachexia. This placebo controlled dose range study will evaluate the safety and efficacy of anamorelin HCl in patients with non-small cell lung cancer, a cancer associated with a high prevalence of cachexia.

ELIGIBILITY:
Inclusion Criteria:

* stage IIIB or IV NSCLC
* eligible for treatment of NSCLC with paclitaxel and carboplatin +/- bevacizumab

Exclusion Criteria:

* mixed large and small cell histologies for lung cancer
* significant obesity, BMI > 30

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 228 (Actual)
Dates: Start 2008-03; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Hand grip strength and body weight | Twelve weeks

SECONDARY OUTCOMES:
Quality of Life and Biomarker | Twelve weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Temel, MD, Study Director — Massachusetts General Hospital
Locations (33):
- United States (19):
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Osler Medical, Melbourne, Florida
  - Augusta Oncology Associates, Augusta, Georgia
  - South Georgia Medical Center, Valdosta, Georgia
  - Investigative Clinical Research of Indiana, Indianapolis, Indiana
  - John Hopkins University, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Center, Boston, Massachusetts
  - Caritas St. Elizabeth's Medical Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - The West Clinic, Corinth, Mississippi
  - The West Clinic, Southaven, Mississippi
  - Washington University School of Medicine, St Louis, Missouri
  - Duke University Medical Center, Durham, North Carolina
  - South Carolina Cancer Specialists, Hilton Head Island, South Carolina
  - The West Clinic, Memphis, Tennessee
  - Baylor College of Medicine/VAMC, Houston, Texas
  - The Methodist Hospital Research Institute, Houston, Texas
  - North West Medical Specialties, PLLC, Puyallup, Washington
- India (14):
  - Regional Cancer Centre Indira Gandhi Institute of Medical Sciences, Patna, Bihar
  - Cancer Clinic 208, Nagpur, Maharashtra
  - Noble Hospital, Pune, Maharashtra
  - Ruby Hall Clinic, Pune, Maharashtra
  - Kaushalya Medical Foundation Trust Hospital, Thane, Maharashtra
  - SEAROC Cancer Center, Jaipur, Rajasthan
  - Jawaharlal Nehru Cancer Hospital and Research Centre, Bhopal
  - Kamakshi Memorial Hospital, Chennai
  - Dharamshila Cancer Hospital and Research Center, Delhi
  - Bhagwan Mahaveer Cancer Hospital and Resaerch Center, Jaipur
  - Birla Cancer Centre SMS Medical College Hospital, Jaipur
  - Kodlikeri Memorial Hospital, Maharashtra
  - Jaslok Hospital and Research Centre, Mumbai
  - Shatabdi Super Speciality Hospital, Mumbai Naka, Nasik